CLINICAL TRIAL: NCT02219919
Title: Changes in Nociceptive Gain Processing After Physical Therapy and Surgery in Carpal Tunnel Syndrome: A Randomized Clinical Trial
Brief Title: Nociceptive Gain Processing After Physical Therapy in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Hospital Universitario Fundación Alcorcón (Other); Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Proffesor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUFA-12/14
Record Dates: First submitted 2014-08-16; First posted 2014-08-19 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Pain; Sensitivity; Pain Thresholds; Sensitization; Physical Therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain; Hypersensitivity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Therapy Group (Experimental): The physical therapy group will receive 3 treatment sessions of manual therapy including desensitization maneuvers of the central nervous system of 30 minutes of duration, once per week.
  Interventions: Other: Physical Therapy Group
- Surgical Group (Active Comparator): The surgical group will receive a surgical procedure consisting of the decompression and release of the median nerve at the carpal tunnel performed by an experienced surgeon according to standardized protocols.
  Interventions: Other: Surgical Group

INTERVENTIONS:
Other: Surgical Group — The surgical group will receive a surgical procedure consisting of the decompression and release of the median nerve at the carpal tunnel performed by an experienced surgeon according to standardized protocols.
  Arms: Surgical Group
Other: Physical Therapy Group — The physical therapy group will receive 3 treatment sessions of manual therapy including desensitization maneuvers of the central nervous system of 30 minutes of duration, once per week.
  Arms: Physical Therapy Group

SUMMARY:
This randomized clinical trial will investigate changes in pain intensity and nociceptive gain processing after the application of either physical therapy or surgery in women with carpal tunnel syndrome (CTS). The purpose of this study will be to determine changes in pain intensity, widespread pressure pain sensitivity and segmental thermal changes after the application of a physical therapy program based on desensitization maneuvers of the central nervous system or endoscopic surgery in women with CTS at medium and long-term follow-up periods. We hypothesize that the physical therapy intervention targeted to desensitization of the central nervous system is more effective than surgical intervention for modulating altered nociceptive gain processing in women with CTS.

DETAILED DESCRIPTION:
There is increasing evidence suggesting that carpal tunnel syndrome (CTS) represents a complex pain syndrome including both peripheral and central sensitization mechanisms. In fact, patients with unilateral CTS exhibit bilateral widespread pressure hyperalgesia and bilateral pain hypersensitivity suggesting the presence of altered nociceptive gain processing. In addition, these sensitization processes seem to be independent of electro-diagnostic findings. Previous studies support the use of physical therapy and surgical interventions for the management of pain and disability in these patients. However, there is no evidence related to changes in nociceptive gain process after the application of any therapeutic intervention. Preliminary evidence suggests that manual therapies can modulate sensitization mechanisms. Therefore, our objective is to conduct a randomized clinical trial to determine if manual therapies including desensitization maneuvers of the central nervous system are effective to decrease widespread pressure pain and thermal pain hypersensitivity in women with CTS.

ELIGIBILITY:
Inclusion Criteria:

* pain and paresthesia in the median nerve distribution
* increasing symptoms during the night,
* positive Tinel sign,
* positive Phalen sign,
* symptoms had to have persisted for at least 6 months
* deficits of sensory and motor median nerve conduction according to guidelines of the American Association of Electrodiagnosis, American Academy of Neurology, and the American Physical Medicine and Rehabilitation Academy

Exclusion Criteria:

* any sensory/motor deficit related to the ulnar or radial nerve;
* older than 65 years of age;
* previous surgical intervention or steroid injections;
* multiple diagnoses of the upper extremity (eg, cervical radiculopathy);
* history of neck, shoulder, or upper limb trauma (whiplash);
* history of a systemic disease causing CTS (eg, diabetes mellitus or thyroid disease);
* history of other medical conditions (eg, rheumatoid arthritis, fibromyalgia);
* pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in widespread pressure pain thresholds between baseline and follow-up periods | Baseline and 3, 6, 9 and 12 months after the intervention.
  Pressure pain thresholds over the median, ulnar and radial nerves, and over the cervical spine, the second metacarpal, and tibialis anterior muscles will be bilaterally assessed.

SECONDARY OUTCOMES:
Changes in heat and cold pain thresholds between baseline and follow-up periods | Baseline and 3, 6, 9 and 12 months after the intervention
  Heat and cold pain thresholds over the carpal tunnel and the thenar eminence will be bilaterally assessed.
Changes in pain intensity between baseline and follow-ups periods | Baseline and 3, 6, 9 and 12 months after the intervention
  An 11-point Numerical Pain Rating Scale (NPRS, 0: no pain - 10: maximum pain) will be used to assess the patients' current level of hand pain and the worst and lowest level of pain experienced in the preceding week. The mean value of the 3 scores will be used in the analysis at each follow-up period.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Fundación Alcorcon, Alcorcón, Madrid
  - Universidad Rey Juan Carlos, Alcorcón, Madrid